CLINICAL TRIAL: NCT06124625
Title: Effects of Rehabilitation Combined With a 12-week Maintenance Program Compared to Rehabilitation Alone in Post-COVID-19 - a Randomized, Controlled Trial.
Brief Title: Effects of Rehabilitation Combined With a Maintenance Program Compared to Rehabilitation Alone in Post-COVID-19
Acronym: ReLoAd2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Bavarian State Ministry of Health and Care (Funding) (Unknown); Deutsche Rentenversicherung (German pension insurance) (Unknown); Betriebskrankenkassen Landesverband Bayern (Bavarian health insurance) (Design) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Head of pulmonology, head of institute for pulmonary rehabilitation research, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Reload 2.0
Record Dates: First submitted 2023-11-08; First posted 2023-11-09 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Post-COVID-19 Syndrome
Keywords: rehabilitation; maintenance program
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rehabilitation maintenance program (Active Comparator)
  Interventions: Procedure: Rehabilitation combined to a digital maintenance program
- No Rehabilitation maintenance program (Placebo Comparator)
  Interventions: Procedure: Rehabilitation without maintenance program

INTERVENTIONS:
Procedure: Rehabilitation combined to a digital maintenance program — Individuals in this group undergo a 3-week inpatient rehabilitation program followed by a 12-week maintenance program (2 sessions per week à 90 minutes, digital and live). The multimodal programs consist of physiotherapy, training therapy, medical support, cognitive training, education and psychological support.
  Arms: Rehabilitation maintenance program
Procedure: Rehabilitation without maintenance program — Individuals in this group undergo a 3-week inpatient rehabilitation program followed by a 12-week usual care period.
  Arms: No Rehabilitation maintenance program

SUMMARY:
Infection with SARS-CoV-2 virus leads to persistent symptoms for more than 12 weeks in 15% of cases ("post-COVID syndrome"). Symptoms like fatigue, dyspnoea, limitations in physical performance and activities, head ache, anxiety symptoms, and depression are heterogenous which limit physical health and participation in daily life activities.

In the last years, multidisciplinary rehabilitation programs showed benefits in quality of life and symptom intensity in patients with post-COVID. Therefore, rehabilitation programs are recommended for individuals with Post-COVID by official sites like the German Society of Pulmonology and the European Respiratory Society.

Own first data (published at the ERS conference 2023) revealed that one the one hand, inpatient rehabilitation is effective, however, on the other hand, it is challenging to maintain these effects after completing the program. Therefore, the aim of this study is to sustain these benefits by using a digital maintenance program following the rehabilitation program compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID-syndrome (Definition WHO)
* Entered the rehabilitation process at the Schoen Klinik Berchtesgadener Land

Exclusion Criteria:

* No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline quality of life assessed by Short-Form 12 questionnaire at week 4 and week 19 | Baseline, week 4, week 19
  The scale of the physical and mental Health component summary score ranges from minimum 0 to maximum 100 points with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Change from baseline post-COVID-related symptoms at week 4 and week 19 | Baseline, week 4, week 19
  The number of COVID-symptoms will recorded as well as their intensity will be rated on a scale from 0 [not relevant] until 10 [very severe symptom].
Change from baseline lung function at week 4 and week 19 | Baseline, week 4, week 19
  following Parameters will be collected:Pimax
Change from baseline fatigue symptoms at week 4 and week 19 | Baseline, week 4, week 19
  Fatigue Assessment Scale will be used
Change from baseline exercise capacity at week 4 and week 19 | Baseline, week 4, week 19
  1-minute sit to stand test will be performed (maximum repetitions of squats in one minute)
Change from baseline physical activity at week 4 and week 19 | Baseline, week 4, week 19
  Activity will be measure in steps per day using a wearable from Polar
Change from baseline quality of life at week 4 and week 19 | Baseline, week 4, week 19
  EQ-5D-5L questionnaire will be used.
Change from the use of health care service at week 4 and week 19 | Baseline, week 4, week 19
  Frequency of therapeutical, medical and psychological sessions will be documented.
Change from the use of medications at week 4 and week 19 | Baseline, week 4, week 19
  Amount and kind of medication will be documented.
Change from rate of sickness at week 4 and week 19 | Baseline, week 4, week 19
  Days of sickness will be documented.
Change from workability at week 4 and week 19 | Baseline, week 4, week 19
  Work ability index will be used
Change from ICF functionality at week 4 and week 19 | Baseline, week 4, week 19
  Indicators of rehabilitation status questionnaire (IRES-3) will be used.
Change from sleep quality at week 4 and week 19 | Baseline, week 4, week 19
  Sleep quality will be assessed by using the Pittsburgh Sleep Quality Index (total score ranges from 0 to 21 with higher scores indicating higher impairment)
Change from depression symptoms at week 4 and week 19 | Baseline, week 4, week 19
  Patient Health Questionnaire 9 will be used. The total score ranges from 0 to 27 points with higher scores indicating worse Depression symptoms
Change from anxiety symptoms at week 4 and week 19 | Baseline, week 4, week 19
  Generalized Anxiety Disorder Scale 7 will be used. The total score ranges from 0 to 21 points with higher scores indicating more anxiety symptoms
Change from resilience at week 4 and week 19 | Baseline, week 4, week 19
  Resilience scale RS-13 will be used.
Change from cognition at week 4 and week 19 | Baseline, week 4, week 19
  Cognition will be measured via the software RehaCom (by Hasomed GmbH).
Change from cognitive impairment at week 4 and week 19 | Baseline, week 4, week 19
  Cognitive impairment will be measured by Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Koczulla, PROF, Principal Investigator — Schön Klinik Berchtesgadener Land
Locations (1):
- Schone Klinik Berchtesgadener Land, Schönau am Königssee, Germany